CLINICAL TRIAL: NCT06666933
Title: Study of Time-restricted Eating (TRE) to Clinical Pregnancy Rate Via IVF/ICSI in Women With PCOS and Glucose Metabolism Disorder: A Multicenter Randomized Controlled Trial (RCT)
Brief Title: Study of Time-restricted Eating (TRE) to Clinical Pregnancy Rate in PCOS Women With Glucose Metabolism Disorder Via IVF/ICSI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Shanghai First Maternity and Infant Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Shengjing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LY2024-160
Record Dates: First submitted 2024-10-20; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: PCOS; Glucose Metabolism Disorder; IVF Outcome
Keywords: PCOS; Glucose Metabolism Disorder; IVF; ICSI; time-restricted eating
MeSH Terms: conditions — Glucose Metabolism Disorders; Intermittent Fasting | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating with metformin (Experimental): TRE (eating is allowed from 8am to 4pm without limitation in calories) with metformin 1g bid po for 6 weeks
  Interventions: Behavioral: Time restricted eating; Drug: Metformin
- Metformin only (Other): Taking metformin 1g bid po for 6 weeks only
  Interventions: Drug: Metformin

INTERVENTIONS:
Behavioral: Time restricted eating — TRE (eating is allowed from 8am to 4pm without limitation in calories) with metformin 1g bid po for 6 weeks
  Arms: Time restricted eating with metformin
Drug: Metformin — Taking metformin 1g bid po only for 6 weeks as control

SUMMARY:
Investigate the effect and mechanism of time-restricted eating (TRE) on the clinical pregnancy rate in women with PCOS and glucose metabolism disorder via IVF/ ICSI.

DETAILED DESCRIPTION:
In this multicenter randomized controlled study, investigators plan to recruit 254 patients, aged 20-38, with PCOS and glucose metabolism disorder. PCOS diagnostic criteria based on Rotterdam 2003 criteria, glucose metabolism disorder are diagnosed by 1998 WHO diagnostic criteria, with HbA1c≤7%. Participants selected are overweight or obese (24Kg/m2 ≤ BMI ≤40Kg/m2), and are planned to start the 1st/ 2nd cycle of IVF/ ICSI.

Investigators divide these patients randomly into 2 groups (each group with 127 patients): metformin only group (control group) and TRE with metformin group. Every participant receives the specific treatment according to the group for at least 6 weeks. During the intervention period, follow-ups, blood chemistry tests and examinations are recorded every 2 weeks. After the intervention period, IVF/ ICSI is carried out. GnRH-agonist- or/and hCG-triggered is used for ovarian stimulation. Ovum retrieval will be carried out 34-36h after ovarian stimulation. Blood hCG is tested after 12-14 days after embryonic transfer. For patients with positive hCG, clinical pregnancy is confirmed by observing gestational sac via transvaginal ultrasound after 4-5 weeks.

Investigators compare the terminal pregnancy-related result and metabolic changes between 2 groups to determine the effect and the possible mechanisms of TRE on IVF/ ICSI clinical pregnancy rate of PCOS with glucose metabolism disorder patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with PCOS based on Rotterdam 2003 (all 3 criteria should be fulfilled);
2. Diagnosed with glucose metabolism disorder (IGT, IFG, IGT with IFG, T2DM) and HbA1c less than or equal to 7%;
3. Age 20-38;
4. Overweight or obese (24Kg/m2 ≤ BMI ≤40Kg/m2);
5. Indication for IVF/ ICSI (repeated ovarian stimulation failure/ Fallopian tube blockage/ male factor) and ready for the 1st/ 2nd cycle of IVF;
6. Cooperative to follow-ups and capable of reporting severe adverse event (SAE);
7. Completed informed consent.

Exclusion Criteria:

1. Unilateral ovary resection;
2. Abnormal uterus cavity (congenital, chronic endometrium inflammation, polyps, adhesion, fibroids, etc);
3. Chromosomal abnormality (either maternal or paternal);
4. Recurrent abortion or recurrent failure of embryo transfer;
5. Metformin allergy/ intolerance;
6. Other serious or uncontrolled diseases (e.g. kidney insufficiency, infection, controlled hypertension, heart disease, etc);
7. Preimplantation genetic testing;
8. Other condition that may impact the results

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 254 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate for the first embryo transfer | 4-5 weeks after the IVF/ ICSI carried out at the end of the 6 weeks intervention
  Clinical pregnancy rate= (number of cycle for 1or more gestational sac is observed via transvaginal ultrasound/ total number of cycle for first embryo transfer)x100%

SECONDARY OUTCOMES:
Number of retrieved oocytes | After the IVF/ ICSI carried out at the end of the 6 weeks intervention
  Includes immature oocytes, mature oocytes and abnormal oocytes from ovum pick-up
Implantation rate | After the IVF/ ICSI carried out at the end of the 6 weeks intervention
  the ration of total number of early gestational sacs to total number of transferred embryos
Abortion rate | After the IVF/ ICSI carried out at the end of the 6 weeks intervention
  the ratio of the number of nonviable pregnancies before 28 weeks of gestation to the number of clinical pregnancies
Number of good quality embryo | After the IVF/ ICSI carried out at the end of the 6 weeks intervention
  Day 3 embryo with 7-9 cells and <10% fragmentation
Weight | From enrollment to the end of treatment at 6 weeks
  Weight change in kg
Fat% | From enrollment to the end of treatment at 6 weeks
  Inbody machine measurement
Lipid profile | From enrollment to the end of treatment at 6 weeks
  Triglycerol, total cholesterol, HDL, LDL, free fatty acid in mmol/L
Blood pressure | From enrollment to the end of treatment at 6 weeks
  Both systolic and diastolic pressure in mmHg
Sex hormone | From enrollment to the end of treatment at 6 weeks
  DHEAs, testosterone, androstadienone, estradiol, LH, FSH, progesterone, prolactin, SHBG
OGTT | From enrollment to the end of treatment at 6 weeks
  Blood glucose level at 0h, 1h, 2h in mmol/L
Insulin stimulation | From enrollment to the end of treatment at 6 weeks
  Serum insulin level at 0h, 1h, 2h in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD, Principal Investigator — RenJi Hospital Department of Endocrinology and Metabolism
Locations (1):
- RenJi Hospital Department of Endocrinology and Metabolism, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided